CLINICAL TRIAL: NCT07248033
Title: Evaluating the Role of Single Photon Emission Computed Tomography/Computed Tomography Derived Quantitative Parameters of Bone Scintigraphy in Characterization of Bone Lesions.
Brief Title: Role of SPECT/CT of Bone Scan in Charactarization of Bone Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: MennaTalla Saber Sabet Mohamed (Other)
Responsible Party: Sponsor-Investigator, MennaTalla Saber Sabet Mohamed, Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: SPECT/CT in bone scan
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Bone Lesions
MeSH Terms: interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SPECT/CT — It is a medical imaging test that combines a Single-Photon Emission Computed Tomography (SPECT) scan with a Computed Tomography (CT) scan to provide both detailed physiological (function) and anatomical (structure) information about the body. A radioactive tracer is injected and detected by the SPECT camera to show organ function, while the CT scan captures precise images of the body's structures, allowing for precise localization of the tracer and identification of abnormalities in a single, comprehensive study.

SUMMARY:
This observational study aims to assess the diagnostic value of SPECT/CT of 99mTc-MDP bone scintigraphy in differentiating begnin from malignant bone lesions. The main question it aims to answer is:

●Can SPECT/CT-derived quantitative parameters (SUVmax, SUVmean) accurately differentiate between begnin and malignant bone lesions in clinical settings? Final diagnostic impression: confirmed by biopsy (if available), or through multidisciplinary radiologic-clinical correlation

DETAILED DESCRIPTION:
Bone lesions represent a common diagnostic challenge in oncology and general radiology, as they may be of malignant, benign, or degenerative origin. Accurate differentiation is essential for guiding appropriate management, avoiding unnecessary biopsies or surgeries, and improving patient outcomes.

Among imaging modalities, 99mTc-methylene diphosphonate (MDP) bone scintigraphy has long been a cornerstone in skeletal evaluation due to its high sensitivity in detecting bone turnover. However, hybrid SPECT/CT imaging, which combines functional and anatomical data, has revolutionized bone imaging by enhancing lesion localization, characterization, and diagnostic specificity.

Recent advances in quantitative SPECT/CT allow the extraction of semi-quantitative parameters, such as the Standardized Uptake Value (SUV), previously limited to PET imaging. These SUV-based parameters have shown promising diagnostic value in distinguishing benign from malignant skeletal lesions.

For instance, SUVmax thresholds derived from 99mTc-MDP SPECT/CT have been proposed in several studies, with malignant lesions often demonstrating higher uptake than benign ones due to increased osteoblastic activity.

In resource-limited settings such as Egypt, access to PET/CT remains constrained due to cost and availability, especially outside major urban centers. Consequently, leveraging the diagnostic utility of quantitative SPECT/CT could bridge the gap in skeletal lesion assessment and aid in earlier detection and treatment planning.

Therefore, this study aims to evaluate the diagnostic value of SPECT/CT-derived SUV in differentiating benign and malignant bone lesions at a tertiary center in Upper Egypt. It will analyze the correlation between SUV metrics, lesion morphology, and final diagnosis, contributing to the growing body of evidence supporting quantitative SPECT/CT in musculoskeletal oncology.

ELIGIBILITY:
Inclusion Criteria:

* Any age referred for 99mTc-MDP SPECT/CT
* Clinical suspicion of either metastatic or degenerative etiology

Exclusion Criteria:

* Case with double malignancies
* Pregnant patients
* Severely ill patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients referred to the Nuclear Medicine Unit at Assiut University, for bone imaging using 99mTc-MDP SPECT/CT due to clinical suspicion of bone lesions.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To measure SUVmax and SUVmean of bone lesions using quantitative SPECT/CT. | Baseline
To compare these values between malignant and degenerative lesions confirmed by clinical, histological, or radiological follow-up. | Baseline

SECONDARY OUTCOMES:
To establish a diagnostic SUV cut-off value that aids in distinguishing between lesion types. | Baseline